CLINICAL TRIAL: NCT00931736
Title: A Randomized Clinical Trial of 4 Months of Rifampin vs. 9 Months of Isoniazid for Latent Tuberculosis Infection. Part 3 - Effectiveness
Brief Title: Randomized Clinical Trial Comparing 4RIF vs. 9INH for LTBI Treatment-effectiveness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Dick Menzies, Director of Respiratory Medicine, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT-94831; ISRCTN05675547 (Other Grant/Funding Number: MCT-94831)
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Latent Tuberculosis Infection
Keywords: Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — Isoniazid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoniazid (Active Comparator): The dosage of the medication is determined according to the weight of the subject. The dose is once per day, in pill format, for a total daily dose of 300mg if subject weighs ≥ 42 kg, otherwise 200 mg. Total duration of treatment is for 9 months.
  Interventions: Drug: Isoniazid
- Rifampin (Active Comparator): The dosage of the medication is determined according to the weight of the subject. The dose is once per day, in pill format, for a total daily dose of 600 mg if the subject weighs ≥ 50 kg, 450 mg if the subject weighs ≥ 36 kg and < 50 kg, otherwise 300 mg for those weighing < 36 kg. Total duration of treatment is for 4 months.
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Isoniazid — The dosage of the medication is determined according to the weight of the subject. The dose is once per day, in pill format, for a total daily dose of 300mg if subject weighs ≥ 42 kg, otherwise 200 mg. Total duration of treatment is for 9 months.
  Arms: Isoniazid
Drug: Rifampin — The dosage of the medication is determined according to the weight of the subject. The dose is once per day, in pill format, for a total daily dose of 600 mg if the subject weighs ≥ 50 kg, 450 mg if the subject weighs ≥ 36 kg and < 50 kg, otherwise 300 mg for those weighing < 36 kg. Total duration of treatment is for 4 months.
  Arms: Rifampin

SUMMARY:
On a global scale, tuberculosis (TB) is the single most important infectious cause of morbidity and mortality. The World Health Organization has estimated that one-third of the entire world's population carries latent TB infection. A key TB control strategy is therapy of latent TB infection (LTBI). The current standard regimen is 9 months of Isoniazid (9INH). This regimen has excellent efficacy if taken regularly, but its effectiveness is substantially reduced by poor compliance. Serious side effects, such as hepato-toxicity can occur. Three shorter alternatives have been recommended: 6 months INH (6INH), 2 months Rifampin - Pyrazinamide (2RIF-PZA) and 4 months Rifampin (4RIF). The regimen of 6INH is less efficacious than 9INH, while 2RIF-PZA has been largely abandoned because of serious toxicity. Based on some evidence in treatment of LTBI, and extrapolating from extensive experience with treatment of active TB, it is believed that 4RIF has similar efficacy as 9INH. Therefore, the investigators are initiating the first multi-site international randomized trial that will compare the effectiveness of 4RIF and 9INH in preventing active tuberculosis.

DETAILED DESCRIPTION:
On a global scale, tuberculosis (TB) is the single most important infectious cause of morbidity and mortality. The World Health Organization has estimated that one-third of the entire world's population carries latent TB infection. Of these 8 million develop active disease, and 2 million die from TB each year. In Canada, and most other industrialized countries, the incidence of TB fell dramatically from 1900 until the late 1970's, but since then decline has slowed, and TB continues to cause significant morbidity, and mortality in disadvantaged populations.

A key TB control strategy is therapy of latent TB infection (LTBI). The current standard regimen is 9 months of Isoniazid (9INH). This regimen has excellent efficacy if taken regularly, but its effectiveness is substantially reduced by poor compliance. Serious side effects, such as hepato-toxicity can occur. Three shorter alternatives have been recommended: 6 months INH (6INH), 2 months Rifampin - Pyrazinamide (2RIF-PZA) and 4 months Rifampin (4RIF). Based on some evidence in treatment of LTBI, and extrapolating from extensive experience with treatment of active TB, it is believed that 4RIF has similar efficacy as 9INH.

The investigators have initiated a research program to evaluate the compliance, safety, costs and effectiveness of 4RIF for the treatment of LTBI. In the initial study of 116 patients, 4RIF was associated with significantly higher completion rates (90% vs 70%). The second phase of this study, conducted in Montreal, Toronto, Kingston, Saskatoon, Calgary, and Edmonton, plus Brazil and Saudi Arabia, compared the rates of serious adverse events (SAE) with the two regimens. These were adjudicated by an independent three member review panel, blinded to study drug. In this phase, among 420 subjects randomized to 4RIF overall rate of Grade 3-4 SAE was 2.4% compared to 5.6% among the 427 taking 9INH (p=.02). Grade 3-4 hepatotoxicity was very significantly lower (0.7% vs 3.8%; p=.003). Health system costs were also significantly lower, and completion rates significantly higher with 4RIF Therefore the conditions have been met to conduct the first randomized trial that will compare effectiveness of 4RIF and 9INH in preventing tuberculosis. Among the moderate to high risk subjects that will be eligible, the anticipated cumulative risk of active TB, if untreated, will be at least 3% during a follow-up of 28 months after randomization. We anticipate 50% completion rate with 9INH, providing an effectiveness of 45% (based on known efficacy of 90%). To detect superior effectiveness of 4RIF, assuming 80% completion, and 10% loss in follow-up, plus accounting for cluster randomization of household contacts we would require enrolment of 3283 subjects per arm, or a total of 6,566 subjects. This is reduced to 5720, because the 847 already randomized in Phase 2, were randomized, treated and followed for 28 months post-randomization to determine occurrence of active TB - using the same methods described in this proposal.We have assumed 4RIF efficacy of 90%, based on available evidence. If 50% of the 2,898 randomized to each group complete therapy and 28 months follow-up, this would provide more than 90% power, to confirm non-inferior efficacy of 4RIF, if the non-inferiority margin was 25% - equivalent to a minimum efficacy of 4RIF of 65%. (In other words, we would declare 4RIF non-inferior to 9INH if the efficacy of 4RIF was not more than 25% worse than 9INH.) This efficacy has been considered sufficient for authoritative recommendations of 6INH, which has had efficacy of 40-69% in trials Eligible consenting subjects will be randomized in equal numbers to 9INH or 4RIF, by a web-based registration and randomization program, stratified by site in blocks of variable size (2-8 subjects). Subjects will be followed by their usual providers during therapy and then every 3 months up to 28 months post-randomization or the occurrence of a study end-point. The primary study outcome is the occurrence, during the 28 months after randomization, of microbiologically or histologically confirmed active TB. The final diagnosis will be based on the majority opinion of an independent 3-member clinical review panel, who will review all subjects investigated for TB, without knowledge of study drug, nor the clinical diagnosis. Planned sub-group analysis will compare rates of active TB in those who complete treatment per protocol (efficacy). Secondary outcomes include occurrence of confirmed plus probable active TB, Grade 3-4 adverse events (judged by another blinded, independent 3-member panel as in Phase 2), occurrence of drug resistant active TB, and costs - from the health system perspective. To accomplish this, in Canada one site has been added in Vancouver, the site in Brazil is doubled, and new sites in Korea, Australia, Indonesia, Benin, Guinea and Ghana (West Africa) have been added.

In addition to the parent trial, the investigators will include an additional component called "the Biomarker Study". For this part of the study the investigators will take an additional 10 mls of blood pre-treatment, as well as at four and nine months after starting treatment. In total an extra 30ml of blood (equal to 2 tablespoons) will be required over 9 months, and two additional veni-punctures, since veni-punctures will not be routinely performed at the 4 and 9 month time points. Three of the 10 ml will be used for the QFT-GIT test, the remaining 7 ml will have the serum separated and stored at -80°C for future biomarker studies. For subjects who were randomized to 4RIF, the blood draw at nine months will require an extra visit to the clinic, for which study subjects will be compensated. No specimens will be stored for future genetic testing. For the present time only the Montreal site will participate in this component. Other sites will join once funding is secured. All lab assays will be performed in the final year of the study, to enhance cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 years and older) with documented positive TST (or in the absence of TST, a documented positive QFT) and prescribed 9 months of Isoniazid for LTBI, following authoritative recommendations.

Exclusion Criteria:

* Patients who were contacts of TB cases known to be resistant to Isoniazid, Rifampin, or both.
* Known HIV-infected individuals on anti-retroviral agents whose efficacy would be substantially reduced by Rifampin, unless therapy can safely be changed to agents not affected by Rifampin.
* Pregnant women - Rifampin and Isoniazid are considered safe in pregnancy but therapy is usually deferred until 2-3 months post-partum to avoid fetal risk and the potential for increased hepato-toxicity immediately post partum.
* Patients on any medication with clinically important drug interactions with Isoniazid or Rifampin, which their physician believes would make either arm contra-indicated.
* Patients with a history of allergy/hypersensitivity to Isoniazid or to Rifampin, Rifabutin or Rifapentine.
* Patients with active TB. Patients initially suspected to have active TB can be randomized once this has been excluded.
* Patients who have already started LTBI therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6031 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Confirmed active TB during 28 months after randomization | 7 years total with data analysis
  Confirmed active TB during 28 months after randomization will be defined as a positive culture for M. tuberculosis, positive Nucleic acid amplification test for M TB complex, or caseating granulomas in a biopsy from any site. Positive AFB smears will be considered false positive if cultures are negative, but will be considered confirmatory, if cultures failed (for example if contamination or other technical problem occurs).

SECONDARY OUTCOMES:
Confirmed active TB in compliant participants | 7 years total with data analysis
  Compare the cumulative incidence of confirmed active TB among those who took at least 80% of doses of the LTBI treatment to which they were randomized, in less than 120% of the allowed time (i.e. efficacy ).
Probable and confirmed active TB | 7 years total with data analysis
  Compare the cumulative incidence of probable, as well as confirmed, active TB between patients randomized to the two regimens during 28 months following randomization.
Rate of Grade 3 & 4 adverse events | 7 years including data analysis
  Compare rates of Grades 3 &4 adverse events during treatment between subjects randomized to the two regimens.
Comparative cost-effectiveness of regimens | 7 years including data analysis
  Compare health system costs, and cost-effectiveness of the two regimens, in the different sites.
Occurrence of drug resistance in confirmed cases of active TB | 7 years including data analysis
  Describe occurrence of drug resistance (to INH or RIF) among subjects who develop confirmed active TB.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Menzies, MD, Principal Investigator — McGill University / McGill University Health Centre
Locations (12):
- Woolcock Institute of Medical Research, Sydney, New South Wales, Australia
- Centre de Pneumophthysiologie, Cotonou, Benin
- Universidade Gama Filho, Centro de Ciências Biológicas e da Saúde, Rio de Janeiro, Brazil
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - British Columbia Centre for Disease Control, Vancouver, British Columbia
  - Montreal Chest Institute, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Research and Development Unit, Komfo Anokye Teaching Hospital, Kumasi, Ghana
- Service de Phtisiologie, Hopital National Ignace Deen, Conakry, Guinea
- Health Research Unit, Faculty of Medicine, Bandung, West Java, Indonesia
- King Fahad National Guard Hospital, Riyadh, Saudi Arabia
- Korean Institute of Tuberculosis, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Allard-Gray A, Boakye I, Camara A, Eisenbeis L, Guimaraes-Teixeira E, Sow O, Zielinski D, Campbell JR, Menzies D. Factors Associated With Discontinuation of Tuberculosis Preventive Treatment: Post Hoc Analysis of 2 Randomized, Controlled Trials. Clin Infect Dis. 2023 Jul 5;77(1):84-93. doi: 10.1093/cid/ciad164. PMID 36949623
- [Derived] Campbell JR, Al-Jahdali H, Bah B, Belo M, Cook VJ, Long R, Schwartzman K, Trajman A, Menzies D. Safety and Efficacy of Rifampin or Isoniazid Among People With Mycobacterium tuberculosis Infection and Living With Human Immunodeficiency Virus or Other Health Conditions: Post Hoc Analysis of 2 Randomized Trials. Clin Infect Dis. 2021 Nov 2;73(9):e3545-e3554. doi: 10.1093/cid/ciaa1169. PMID 32785709
- [Derived] Bastos ML, Campbell JR, Oxlade O, Adjobimey M, Trajman A, Ruslami R, Kim HJ, Baah JO, Toelle BG, Long R, Hoeppner V, Elwood K, Al-Jahdali H, Apriani L, Benedetti A, Schwartzman K, Menzies D. Health System Costs of Treating Latent Tuberculosis Infection With Four Months of Rifampin Versus Nine Months of Isoniazid in Different Settings. Ann Intern Med. 2020 Aug 4;173(3):169-178. doi: 10.7326/M19-3741. Epub 2020 Jun 16. PMID 32539440
- [Derived] Campbell JR, Trajman A, Cook VJ, Johnston JC, Adjobimey M, Ruslami R, Eisenbeis L, Fregonese F, Valiquette C, Benedetti A, Menzies D. Adverse events in adults with latent tuberculosis infection receiving daily rifampicin or isoniazid: post-hoc safety analysis of two randomised controlled trials. Lancet Infect Dis. 2020 Mar;20(3):318-329. doi: 10.1016/S1473-3099(19)30575-4. Epub 2019 Dec 19. PMID 31866327
- [Derived] Menzies D, Adjobimey M, Ruslami R, Trajman A, Sow O, Kim H, Obeng Baah J, Marks GB, Long R, Hoeppner V, Elwood K, Al-Jahdali H, Gninafon M, Apriani L, Koesoemadinata RC, Kritski A, Rolla V, Bah B, Camara A, Boakye I, Cook VJ, Goldberg H, Valiquette C, Hornby K, Dion MJ, Li PZ, Hill PC, Schwartzman K, Benedetti A. Four Months of Rifampin or Nine Months of Isoniazid for Latent Tuberculosis in Adults. N Engl J Med. 2018 Aug 2;379(5):440-453. doi: 10.1056/NEJMoa1714283. PMID 30067931